CLINICAL TRIAL: NCT00000770
Title: A Comparative Study of a Combination of Zidovudine, Didanosine, and Double-Blinded Nevirapine Versus a Combination of Zidovudine and Didanosine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 241; 11218 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nevirapine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To assess the safety and toxicity of zidovudine (AZT)/didanosine (ddI) versus AZT/ddI combined with nevirapine in HIV-infected patients, and to obtain preliminary anti-HIV activity data using immunologic and virologic markers.

Previous in vitro studies suggest that HIV that has already developed resistance to AZT and ddI is less able to develop resistance to nevirapine, a non-nucleoside reverse transcriptase inhibitor. Thus, convergent combination therapy with these three drugs in HIV-infected patients may prove more effective.

DETAILED DESCRIPTION:
Previous in vitro studies suggest that HIV that has already developed resistance to AZT and ddI is less able to develop resistance to nevirapine, a non-nucleoside reverse transcriptase inhibitor. Thus, convergent combination therapy with these three drugs in HIV-infected patients may prove more effective.

Patients are randomized to receive AZT/ddI plus either nevirapine or placebo daily for 48 weeks, with possible extension for at least 12 weeks. At eight participating sites, ACTG 808 and 809 will be conducted as virologic and pharmacokinetic substudies.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis for patients with CD4 count < 200 cells/mm3 or a prior history of PCP.

Allowed:

* Trimethoprim with sulfamethoxazole or dapsone, intravenous pentamidine, atovaquone, primaquine-clindamycin or trimetrexate for acute PCP.
* Topical antifungals, clotrimazole, ketoconazole, fluconazole, and amphotericin B for treatment of mucosal and esophageal candidiasis.
* Prophylaxis or therapy for opportunistic infections, as indicated, with other medications such as itraconazole, isoniazid, pyrazinamide, clofazimine, clarithromycin, azithromycin, ethambutol, amikacin, ciprofloxacin, ofloxacin, pyrimethamine, sulfadiazine, and clindamycin.
* Maintenance therapy for opportunistic infections as long as patients have been on a stable dosage regimen for 1 month prior to study entry.
* Ganciclovir for CMV retinitis or gastrointestinal disease as long as patients have been on a stable dose for at least 1 month prior to study entry with no grade 3 or 4 neutropenia or dependence on G-CSF.
* Acyclovir (<= 1000 mg/day) for maintenance of herpes simplex virus infections.
* Erythropoietin or G-CSF if clinically indicated.
* Antibiotics for bacterial infections unless specifically excluded.
* Rifampin or rifabutin.
* Symptomatic treatments such as antipyretics, analgesics, and antiemetics.

Concurrent Treatment:

Allowed:

* Local radiation therapy.

Prior Medication: Required:

* At least 6 months of prior cumulative nucleoside therapy with AZT, ddI, or ddC, given as monotherapy or in combination.

Patients must have:

* Prior or current documentation of HIV seropositivity by ELISA confirmed by Western blot, positive HIV antigen, or positive HIV culture, or a second antibody test by a method other than ELISA.
* CD4 count <= 350 cells/mm3.
* Prior cumulative nucleoside therapy of >= 6 months.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Antiretroviral therapies other than study medications.
* Systemic corticosteroids given consecutively for > 21 days.
* Induction or maintenance with foscarnet.
* Systemic cytotoxic chemotherapy for a malignancy.
* Erythromycin.
* Coumadin/warfarin.
* Phenytoin or phenobarbital.
* Amoxicillin/clavulanate acid (Augmentin) or ticarcillin/clavulanate acid (Timentin).

Patients with the following prior conditions are excluded:

* History of pancreatitis.
* History of intolerance to 500 or 600 mg/day AZT or to 400 mg/day ddI tablets or 500 mg/day ddI sachets.
* History of grade 2 or worse peripheral neuropathy.

Prior Medication:

Excluded at any time:

Prior non-nucleoside reverse transcriptase inhibitors (NVP; L697,611; TIBO; atevirdine).

Excluded within 14 days prior to study entry:

* Acute treatment for a serious infection or any opportunistic infection.
* Biologic response modifiers such as interferon and IL-2.
* Erythromycin.
* Coumadin/warfarin.
* Phenytoin or phenobarbital.
* Ticarcillin/clavulanate acid (Timentin) or amoxicillin/clavulanate acid (Augmentin).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Study Completion 1994-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D'Aquila R, Study Chair; Hirsch M, Study Chair
Locations (44):
- United States (44):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - Summitt Med Ctr / San Francisco Gen Hosp, Oakland, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Comprehensive Health Care Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Samaritan Village Inc / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Wake County Dept of Health, Raleigh, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Girard Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania

REFERENCES:
- [Background] D'Aquila RT, Hughes MD, Johnson VA, Fischl MA, Sommadossi JP, Liou SH, Timpone J, Myers M, Basgoz N, Niu M, Hirsch MS. Nevirapine, zidovudine, and didanosine compared with zidovudine and didanosine in patients with HIV-1 infection. A randomized, double-blind, placebo-controlled trial. National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group Protocol 241 Investigators. Ann Intern Med. 1996 Jun 15;124(12):1019-30. doi: 10.7326/0003-4819-124-12-199606150-00001. PMID 8633815
- [Background] Dusek A, Hall D, Lamson M, Myers M. Once-daily dosing of nevirapine: a retrospective, cross-study analysis. Int Conf AIDS. 1998;12:85 (abstract no 12360)
- [Background] Leigh Brown AJ, D'Aquila RT, Johnson VA, Kuritzkes DR, Richman DD. Baseline sequence clusters predict response to combination therapy in ACTG 241. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:211 (abstract no 704)
- [Background] Fiscus SA, Welles SL, Spector SA, Lathey JL. Length of incubation time for human immunodeficiency virus cultures. J Clin Microbiol. 1995 Jan;33(1):246-7. doi: 10.1128/jcm.33.1.246-247.1995. PMID 7699053
- [Background] D'Aquila RT, Sutton L, Savara A, Hughes MD, Johnson VA. CCR5/delta(ccr5) heterozygosity: a selective pressure for the syncytium-inducing human immunodeficiency virus type 1 phenotype. NIAID AIDS Clinical Trials Group Protocol 241 Virology Team. J Infect Dis. 1998 Jun;177(6):1549-53. doi: 10.1086/515307. PMID 9607832
- [Background] Virus sidesteps convergent therapy. GMHC Treat Issues. 1995 Jan;9(1):6. PMID 11367380
- [Background] Precious H, Leigh Brown AJ, Gunthard HF, Wong JK, D'Aquila RT, Johnson VA, Kuritzkes DR, Richman DD. A multiple regression model predicting response to combination therapy from baseline sequence data identifies amino acid sites not previously associated with resistance. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:69 (abstract no 14)
- [Background] Zhou XJ, Sheiner LB, D'Aquila RT, Hughes MD, Hirsch MS, Fischl MA, Johnson VA, Myers M, Sommadossi JP. Population pharmacokinetics of nevirapine, zidovudine, and didanosine in human immunodeficiency virus-infected patients. The National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group Protocol 241 Investigators. Antimicrob Agents Chemother. 1999 Jan;43(1):121-8. doi: 10.1128/AAC.43.1.121. PMID 9869576
- [Background] Hall D, Robinson P, Cort S, Kohlbrenner V, Leitz G, Myers M. Duration of effect of nevirapine (NVP), a cross-trial analysis of three controlled studies. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:79
- [Background] Hughes MD, Johnson VA, Hirsch MS, Bremer JW, Elbeik T, Erice A, Kuritzkes DR, Scott WA, Spector SA, Basgoz N, Fischl MA, D'Aquila RT. Monitoring plasma HIV-1 RNA levels in addition to CD4+ lymphocyte count improves assessment of antiretroviral therapeutic response. ACTG 241 Protocol Virology Substudy Team. Ann Intern Med. 1997 Jun 15;126(12):929-38. doi: 10.7326/0003-4819-126-12-199706150-00001. PMID 9182469